CLINICAL TRIAL: NCT06120426
Title: En Bloc Resection Versus Separation Surgery Combined With Radiotherapy for the Treatment of Spinal Oligometastatic Tumor-A Multi-center, Prospective, Randomized, Controlled Study.
Brief Title: En Bloc Resection Versus Separation Surgery Combined With Radiotherapy for the Treatment of Spinal Oligometastatic Tumor.
Status: Recruiting | Type: Observational
Sponsor: Shanghai Changzheng Hospital (Other)
Collaborators: Peking University Third Hospital (Other); Peking University People's Hospital (Other); Henan Cancer Hospital (Other Government); First Affiliated Hospital, Sun Yat-Sen University (Other); Sun Yat-sen University (Other); Zhejiang University (Other); Tianjin Hospital (Other); The First Affiliated Hospital of Nanchang University (Other); The Third Affiliated Hospital of Southern Medical University (Other Government)
Responsible Party: Principal Investigator, Jianru Xiao, shanghaiczh, Shanghai Changzheng Hospital
Other Study IDs: 2023SL050
Record Dates: First submitted 2023-11-02; First posted 2023-11-07 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Spinal Metastases; Spinal Tumor; Radiotherapy; Malignant Bone Tumor; Surgery
Keywords: Total enbloc spondylectomy; Oligometastases
MeSH Terms: conditions — Spinal Cord Neoplasms; Bone Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Total en bloc spondylectomy for spinal oligometastases: Based on the medical history, physical signs, and imaging examination results, a definitely diagnosis of spinal oligometastasis tumor was made and perform a Total en bloc spondylectomy.
  Interventions: Procedure: total en bloc spondylectomy
- Separation surgery combined with radiotherapy for spinal oligometastases: Based on the medical history, physical signs, and imaging examination results, a definitely diagnosis of spinal oligometastasis tumor was made and perform a Separation surgery. After surgical recovery, take a radiotherapy.

INTERVENTIONS:
Procedure: total en bloc spondylectomy — Total enbloc resection (TES) is one of the most challenging surgeries in spinal surgery and a classic surgical method. It not only relieve spinal cord compression and delays tumor recurrence, but also prolongs patient survival, significantly reduces hand surgery trauma, and improves surgical safety. However, for cases with extensive tumor invasion, methods such as separation surgery should be used to relieve spinal cord nerve compression, rebuild spinal stability, and provide conditions for postoperative radiotherapy.
  Groups: Total en bloc spondylectomy for spinal oligometastases

SUMMARY:
The purpose of this clinical trial is to explore the impact of En bloc surgery and separation surgery combined with radiation therapy on the prognosis and survival of patients with spinal oligometastatic cancer, describe the clinical results, and optimize future treatment goals

DETAILED DESCRIPTION:
Patients with oligometastatic diseases have been shown to have better prognosis than those with multiple metastatic diseases, and some patients have achieved long-term survival, thus being considered to benefit from more aggressive treatment. Active local treatment, including surgery and/or targeted radiotherapy, such as Stereotactic Radiosurgery (SRS) and Stereotactic body radiotherapy (SBRT), can be performed before or after systemic treatment. For both primary and oligometastatic tumors, radical treatment should be considered in order to achieve better survival and prognosis. The current research has explored the different effects of oligometastatic disease status on the prognosis of various cancers. However, there is currently no clear clinical or experimental confirmation of the impact on the survival and treatment outcomes of patients with oligometastatic spinal cancer. The purpose of this clinical trial is to explore the impact of En bloc hand surgery and separation surgery combined with radiotherapy on the prognosis and survival of patients with oligometastatic spinal cancer, Describe clinical outcomes and optimize future treatment goals

ELIGIBILITY:
Inclusion Criteria:

* 1) Be able to sign written informed consent.
* 2) Age range from 18 to 75 years old, regardless of gender.
* 3) Within conservative treatment, the patient still has uncontrollable pain, metastatic cancer lesions that still progress, spinal instability/potential instability, or symptoms of spinal cord/nerve compression.
* 4) After the patient underwent Positron Emission Tomography-Computed Tomography (PET-CT) examination, it was indicated that there were no more than 3 metastatic organs and no more than 5 metastatic lesions in the whole body of cancer. Among them, there was at least 1 spinal metastasis and at most 5 spinal metastases.
* 5) Imaging examinations (enhanced MRI, enhanced CT, X-ray) indicate the presence of spinal metastasis.
* 6) The expected survival period is ≥ 6 months.
* 7)No other surgical contraindications

Exclusion Criteria:

* 1) Primary tumors of the spine or multiple tumors of the body, with>3 metastatic organs and>5 metastatic sites.
* 2) Previously underwent spinal surgery, or received radiotherapy for the responsible segment of this treatment.
* 3) Severe heart, lung, liver, kidney or other diseases affecting the surgery.
* 4) Having cognitive impairment, sensory aphasia, and inability to understand basic instructions.
* 5) Participated in clinical trials of other drugs or medical devices within 3 months prior to enrollment.
* 6) Infectious diseases.
* 7) Refuse to follow up or participate.
* 8) The researchers determine that the patients are not suitable for enrollment this clinical trail.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: According to the literature results, the median survival period of the experimental group was 20 months, while the median survival period of the control group was 11 months. The total study duration (enrollment+follow-up) was 48 months, and the enrollment time (assuming uniform enrollment speed) was 24 months. The bilateral alpha was 0.05, the beta was 0.2, and the ratio of sample size between the two groups was 2 (experimental group: control group). Through the difference test of median survival time, the experimental sample size was calculated: 110 cases in the experimental group, 55 cases in the control group, a total of 165 cases, Considering 10% detachment, a total of 182 samples are required.
Sampling Method: Probability Sample
Enrollment: 182 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Overall Survival(OS) | after surgery until death due to primary disease or responsible segment
  On the basis of maintaining systemic treatment, compare the overall survival period of En bloc surgery and separation surgery combined with radiation therapy for patients with spinal oligometastatic cancer, after surgery until death due to primary disease or responsible segment.

SECONDARY OUTCOMES:
Local Control Rate(LRC) | a 20% increase in the total diameter of the target lesion observed on imaging from the beginning of the patient's current treatment to baseline.
  Based on the Response Evaluation Criteria in Solid Tumors 1.1 (RECIST 1.1), it is defined as a 20% increase in the total diameter of the target lesion observed on imaging from the beginning of the patient's current treatment to baseline.
Progression-Free Survival(PFS) | The period between the patient receiving this treatment and observing local progression or death from any cause.
  The period between the patient receiving this treatment and observing local progression or death from any cause. Based on the changes in patient imaging and neurological function, comprehensively evaluate whether the local lesion of the spine is progressing.
Brief Pain inventory | 1 day before surgery, 2 weeks after surgery, 1 month after surgery, 3 months after surgery, 6 months after surgery, and 12 months after surgery.
  Use the Brief Pain Inventory (BPI) to score the pain levels 1 day before surgery, 2 weeks after surgery, 1 month after surgery, 3 months after surgery, 6 months after surgery, and 12 months after surgery.
EORTC Quality of Life Questionnaire - Core 30 | 1 day before surgery, 2 weeks after surgery, 1 month after surgery, 3 months after surgery, 6 months after surgery, and 12 months after surgery
  Evaluate the quality of life of patients 1 day before surgery, 2 weeks after surgery, 1 month after surgery, 3 months after surgery, 6 months after surgery, and 12 months after surgery using EORTC Quality of Life Questionnaire - Core 30
Complication | 1 month, 3 months, 6 months, and 12 months after surgery.
  The incidence of vertebral compression fractures: X-ray examination of the surgical area was performed on the first day, within 3 months, within 6 months, and within 12 months respectively.
  Wound complications: Erythrocyte Sedimentation Rate (ESR) and C-reactive protein tests were performed on the first day after surgery. Observe and record the incidence of incision infection, incision non healing, and the need for debridement within 1 month after surgery.
  Other complications: Observe whether the patient experiences bleeding, pulmonary infection, or pulmonary embolism within one month after treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Changzheng hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Result] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Result] Barzilai O, Laufer I, Yamada Y, Higginson DS, Schmitt AM, Lis E, Bilsky MH. Integrating Evidence-Based Medicine for Treatment of Spinal Metastases Into a Decision Framework: Neurologic, Oncologic, Mechanicals Stability, and Systemic Disease. J Clin Oncol. 2017 Jul 20;35(21):2419-2427. doi: 10.1200/JCO.2017.72.7362. Epub 2017 Jun 22. PMID 28640703
- [Result] Barzilai O, McLaughlin L, Amato MK, Reiner AS, Ogilvie SQ, Lis E, Yamada Y, Bilsky MH, Laufer I. Predictors of quality of life improvement after surgery for metastatic tumors of the spine: prospective cohort study. Spine J. 2018 Jul;18(7):1109-1115. doi: 10.1016/j.spinee.2017.10.070. Epub 2017 Nov 6. PMID 29122701
- [Result] Chang JH, Shin JH, Yamada YJ, Mesfin A, Fehlings MG, Rhines LD, Sahgal A. Stereotactic Body Radiotherapy for Spinal Metastases: What are the Risks and How Do We Minimize Them? Spine (Phila Pa 1976). 2016 Oct 15;41 Suppl 20(Suppl 20):S238-S245. doi: 10.1097/BRS.0000000000001823. PMID 27488294
- [Result] Kumar N, Madhu S, Bohra H, Pandita N, Wang SSY, Lopez KG, Tan JH, Vellayappan BA. Is there an optimal timing between radiotherapy and surgery to reduce wound complications in metastatic spine disease? A systematic review. Eur Spine J. 2020 Dec;29(12):3080-3115. doi: 10.1007/s00586-020-06478-5. Epub 2020 Jun 15. PMID 32556627
- [Result] Goetz MP, Callstrom MR, Charboneau JW, Farrell MA, Maus TP, Welch TJ, Wong GY, Sloan JA, Novotny PJ, Petersen IA, Beres RA, Regge D, Capanna R, Saker MB, Gronemeyer DH, Gevargez A, Ahrar K, Choti MA, de Baere TJ, Rubin J. Percutaneous image-guided radiofrequency ablation of painful metastases involving bone: a multicenter study. J Clin Oncol. 2004 Jan 15;22(2):300-6. doi: 10.1200/JCO.2004.03.097. PMID 14722039
- [Result] Dupuy DE, Liu D, Hartfeil D, Hanna L, Blume JD, Ahrar K, Lopez R, Safran H, DiPetrillo T. Percutaneous radiofrequency ablation of painful osseous metastases: a multicenter American College of Radiology Imaging Network trial. Cancer. 2010 Feb 15;116(4):989-97. doi: 10.1002/cncr.24837. PMID 20041484
- [Result] Murali N, Turmezei T, Bhatti S, Patel P, Marshall T, Smith T. What is the effectiveness of radiofrequency ablation in the management of patients with spinal metastases? A systematic review and meta-analysis. J Orthop Surg Res. 2021 Nov 6;16(1):659. doi: 10.1186/s13018-021-02775-x. PMID 34742319
- [Result] D'Souza M, Gendreau J, Feng A, Kim LH, Ho AL, Veeravagu A. Robotic-Assisted Spine Surgery: History, Efficacy, Cost, And Future Trends. Robot Surg. 2019 Nov 7;6:9-23. doi: 10.2147/RSRR.S190720. eCollection 2019. PMID 31807602
- [Result] Kaoudi A, Capel C, Chenin L, Peltier J, Lefranc M. Robot-Assisted Radiofrequency Ablation of a Sacral S1-S2 Aggressive Hemangioma. World Neurosurg. 2018 Aug;116:226-229. doi: 10.1016/j.wneu.2018.05.060. Epub 2018 May 17. PMID 29777897